CLINICAL TRIAL: NCT07221201
Title: Reducing the Intersecting Stigmas of HIV, Violence Victimization, and Mental Health: a Randomized Controlled Pilot Integrating Project YES! Youth Engaging for Success With WHO-Endorsed Mental Health Approaches Among Youth Living With HIV in Ndola, Zambia
Brief Title: Integrating Project YES! With WHO-Endorsed Mental Health Approaches Among Youth Living With HIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); Arthur Davison Children's Hospital (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00024597; 5R01TW012411-03 (NIH)
Record Dates: First submitted 2025-10-24; First posted 2025-10-27 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: HIV - Human Immunodeficiency Virus; Mental Health; Anxiety; Depression in Adolescence; Stigma
Keywords: HIV; Adolescents; Caregivers; Africa; Youth; Intervention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Psychological Well-Being; Anxiety Disorders; Social Stigma

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (Individual Level)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): The comparison group will receive the standard of care. Standard of care at ADCH includes an optional monthly AYALHIV youth group. The comparison arm participants will also be offered referrals to health care providers if they screen positive for depression or have experienced severe forms of violence (a process the investigators utilized and refined during the Project YES! study).
- Project YES+ intervention arm (Experimental): Project YES+ will be about 4 months and will consist of an orientation meeting with the youth client, their caregiver, the healthcare worker and the youth peer mentor to introduce the intervention. Youth clients will then meet with their YPM individually and in groups with other youth living with HIV in the intervention, and go through the WHO- Self Help plus group meetings. Caregivers will also attend three different caregiver group meetings. At the end, there will be a transition group meeting with youth and caregivers together, followed by one last individual mentoring meeting with the youth. All individual and group meetings are facilitated by the youth peer mentor. Study team members will provide reminder calls for youth and their caregivers before intervention meetings and data collection points.
  Interventions: Behavioral: Project YES+ intervention arm

INTERVENTIONS:
Behavioral: Project YES+ intervention arm — Project YES+ integrates Project YES!
  Arms: Project YES+ intervention arm

SUMMARY:
The proposed study will address the intersecting stigmas of HIV, violence and depression among adolescents and young adults (15-24) living with HIV (AYALHIV) in Zambia. The study will integrate a WHO-endorsed mental health approach into an existing HIV-stigma-reducing intervention, and refine measures of internalized and intersecting stigmas, to create and test the feasibility of Project YES+- a combined youth peer mentoring and lay mental health intervention. This research aims to shift HIV care and treatment for AYALHIV by addressing the multiple internalized and intersecting stigmas that impeded antiretroviral adherence and HIV viral suppression.

DETAILED DESCRIPTION:
Nine out of ten AIDS-related deaths among adolescents occur in sub-Saharan Africa (SSA). Despite advances in antiretroviral combination therapy (ART), AIDS-related mortality among adolescents has only decreased 33% since 2010, compared to 66% among children. This slow decline in adolescent deaths is attributed in part to incomplete adherence to ART and subsequent viral failure. Only an estimated 34% of AYALHIV in Zambia, ages 15-24 years, have achieved viral suppression (<1000 copies/mL).

Stigma is increasingly recognized as a modifiable factor impacting ART adherence and viral suppression. Stigma as defined by Goffman is the social devaluation of a person due to an attribute discredited by society, with Parker and Aggleton critically examining stigma as a tool that reinforces inequalities. Different frameworks, such as the mental illness stigma framework and the HIV stigma framework, further delineate stigma into mechanisms experienced by people without the attribute, with the mechanisms being stereotypes, discrimination, and prejudice leading to social rejection, and those with the attribute, with the mechanisms being enacted (experienced), anticipated (beliefs about how others will treat you) and internalized stigma (accepting negative views and devaluing one's self) impacting physical, mental and social health. In this proposed research the investigators focus on internalized HIV stigma among AYALHIV, as well as internalized stigma related to the prevalent youth experiences of violence and depression. Further, the investigators also focus on intersectional stigma, capturing anticipated stigma associated with the complex reality of AYALHIV's multiple social identities instead of one specific attribute. This focus responds directly to this RFA and priority NIH/NIMH future directions for stigma-related research. Evidence shows that internalized stigma is related to viral failure and ART adherence among adults in SSA. Systematic review articles have also examined HIV-internalized stigma interventions; however, a 2019 systematic review of HIV self-stigma interventions in low- and middle-income countries found only one youth focused study from Thailand. In a more recent narrative review, two articles were AYALHIV specific, with only one measuring internalized stigma. In response to this distinct gap in stigma-reducing interventions, and informed by our team's preliminary studies, the investigators developed and tested Project YES! Youth Engaging for Success, to address internalized stigma and HIV outcomes among AYALHIV.

Project YES! is a peer-led facility-based youth mentoring program and is the only CDC evidence-based intervention (EBI) developed in SSA that reduced HIV-internalized stigma among AYALHIV ages 15-24. This RCT found that peer mentoring versus standard of care (SOC) decreased the relative odds of HIV-related internalized stigma (feelings of shame, guilt and worthlessness) by a factor of 0.39 (95% CI:0.21,0.73).) In a stratified analysis, intervention versus SOC participants from a pediatric clinic had a relative increase in the odds of viral suppression (VS) by a factor of 4.7 (95% CI:1.84, 11.78). However, study data also highlighted critical intervention gaps: 74% of AYALHIV experienced physical, sexual and/or emotional violence in the past year, with those experiencing violence at greater risk of viral failure (see preliminary studies).(17) Additionally, AYALHIV who screened positive for depression were less likely to achieve VS (53% vs 62%). Research among South African AYALHIV identified significant, multidirectional pathways linking HIV status and internalized stigma through violence victimization, depression and anticipated stigma, and mental health research clearly links internalized stigma with depression. Few studies, however, examined the relationship between internalized stigma and HIV outcomes, with one finding the impact of discrimination on reduced HIV care retention heightened by internalized stigma. With an estimated 25% of AYALHIV experiencing depression, and the high levels of violence in this population, the investigators must effectively intervene on these pathways to improve HIV outcomes during a developmental stage when youth are "developing and consolidating their sense of self".

To address these gaps the investigators propose integrating WHO-endorsed and lay delivered mental health approaches (e.g. PM+, SH+ and EASE) into our peer mentoring EBI (Project YES!) to create and test Project YES+. The World Health Organization, has various psychological management programs to address mental health conditions through lay workers. Examples of these mental health approaches include Project Management Plus (PM+) and Self Help+, both designed for adults 18+ years, and the Early Adolescent Skills for Emotions (EASE) program designed for young adolescents 10-14 years. While efficacious, the targeted age groups leave a clear gap in service options for 15-19 year olds. By adapting and integrating these mental health approaches into Project YES+, the investigators will specifically provide AYALHIV with problem-management skills through lay peer mentors shown to reduce depression and anxiety. The investigators hypothesize that Project YES+ will also reduce related internalized and intersecting stigmas and improve HIV outcomes. Our refinement of stigma measures will also advance the field's ability to test stigma-reducing interventions to disrupt the pathways among violence, depression, internalized stigma and HIV-related health outcomes. This proposed research will contribute to the field of HIV empirical research and care practices by refining measures and pilot testing a feasible peer led intervention designed to reduce stigma and achieve undetectable viral loads among AYALHIV 15-24 years of age.

STUDY DESIGN The development and pilot testing of Project YES+ will occur in two phases. Phase one has been completed and addressed Aim 1: to integrate an adapted WHO endorsed mental health intervention into Project YES! and Aim 2: to refine stigma measures. To achieve aim 1 the study team first worked with WHO to identify the most promising packages and components to adapt (e.g. PM+, SH+, EASE). After honing in on the key approaches, the investigators then held co-design workshops with AYA and caregivers to refine the Project YES+ To achieve Aim 2, to refine stigma measures, the team conducted cognitive interviewing with youth and caregivers. This phase 1 produced: 1) an age-and-culturally relevant AYALHIV stigma reduction intervention linked to mental health and HIV outcomes, and 2) adapted measures of intersectional, violence-, and depression-related stigmas for AYALHIV.

Phase two is the focus of this registration with clinicaltrials.gov. For phase two, the study team will address Aim 3: to pilot test the intervention, collecting pilot Project YES+ outcomes by conducting an RCT with 50 intervention and 50 comparison AYALHIV and their caregivers who attend HIV care at the Arthur Davison Children's Hospital (ADCH) in Ndola, Zambia (expanding to other clinics if needed to reach the sample size). Individual-level AYA study measures, including stigma, depression, violence, ART adherence, and blood draws for viral testing, will occur at baseline and endline. This data will advance our knowledge on stigma measures and the integration of mental health care in an effective HIV stigma reducing intervention to address the bi-directional associations among HIV, depression, violence victimization, and various internalized stigmas. This data will provide the foundation for a future impact study of Project YES+ on AYALHIV stigmas and HIV outcomes. The specific aim 3 is detailed below:

Aim 3: The purpose of Aim 3 is to test the feasibility of conducting Project YES+ among AYALHIV to prepare preliminary evidence and working knowledge to test the intervention impact in the future. To assess whether 90% of AYAHLIV will attend at least 80% of the intervention sessions with a 90% confidence interval and a margin of error + 10, the investigators will need a minimum sample size of 25 AYALHIV in each study arm. A group sample size of 50 though, will allow us to achieve 74% power to detect a two-sided difference with an alpha of 0.05 of 25 points between the two groups on internalized stigma related to HIV, violence or depression. The investigators know from Project YES! data that a reduction of this size in HIV-internalized stigma is possible. In addition, this sample size will provide valuable data on the proportion of participants reducing psychological distress. At baseline 100% of all AYALHIV participants will have have a positive screen for the Kessler 6 measure of psychological distress and the investigators assume some variability in the proportion with a positive Kessler 6 score in the control group at endline. Group sizes of 50 will achieve 80% power to detect a 20% difference in the Kessler 6 from 95% to 75% between the control and intervention group for a two-sided comparison with alpha=0.05.

ELIGIBILITY:
Inclusion Criteria:

For youth

* Be between ages 15-21
* living within 30-minutes, by personal transportation, of the clinic by self-report,
* and being available to attend sessions and data collection over a 4-8 month time period On ART for at least 6 months
* On first-line ART
* Speaks Bemba

For caregivers

* Being 25 years of age or older
* Caring for an AYALHIV who meets the study eligibility criteria
* Speaks Bemba
* Living within 30-minutes, by personal transportation, of the clinic by self-report
* Being available to attend sessions and data collection over a 4-8 month time period

Exclusion Criteria:

For youth,

* only one youth per household may join.
* Also participants will be excluded from joining the RCT if they are at imminent risk of suicide based on WHO guidance on the Self Help plus program.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-10-25 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of intervention as assessed by percentage of sessions attended | Up to 4 months
  Feasibility of 90% of AYAHLIV attending at least 80% of the intervention sessions with a 90% confidence interval and a margin of error + 10.
Number of intervention participants who report they would recommend Project YES+ to their peers | up to 4 months
  The endline question is "Overall, you would recommend/not recommend this program to another youth living with HIV" with the response options would recommend, would not recomment, decline to answer"
Number of intervention participants who would recommend Project YES+ for caregivers | up to four months
  This outcome will be assessed during endline with the question "Overall, you would recommend/not recommend this program to a caregiver of a another youth living with HIV"

SECONDARY OUTCOMES:
Number of youth participants with a positive composite score consisting of psychological distress (Kessler 6) and one positive stigma score (internalized, violence, mental health and intersectional stigma). | Baseline up to approximately 4 months
  The scales for youth are defined as follows: Kessler 6 measures psychological distress with 6 items and a 4 point likert scale (none of the time to all of the time, 0-24 higher score indicates more psychological distress). Internalized stigma is a 3 point self-stigma scale, with yes/no responses (range is 0-3, higher score indicates more self-stigma). Violence is from the adapted IPV stigma scale that has 19 scale items and a 4 point likert response (disagree alot to agree a lot, 0-76 range with a higher score indicating more violence related stigma). An adapted self-stigma of depression scale consists of 15 items and a 4-point likert scale (disagree alot to agree a lot, 0-60 range, with higher scores indicating more depression related stigma). The adapated intersectional anticipated stigma scale from the intersectional discrimination index and has 9 items and a 4-point likert response (disagree alot to agree a lot, 0-36 range, higher scores indicating more stigma).

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Denison, PhD, Principal Investigator — JHBSPH; Sam Miti, BSc HB, MBcHB, MeMMed-PEDS, Study Director — Arthur Davison Children's Hospital
Locations (1):
- Arthur Davison Children's Hospital, Ndola, Copperbelt, Zambia

IPD SHARING:
Plan to Share IPD: Yes
The investigators will deposit data into an existing data repository for future research. After the study is completed, the de-identified, archived data will be transmitted to and stored in a Data Repository determined in consultation with the NIH Program Officer, for use by other researchers including those outside of the study. Blood samples will not be stored for future research purposes. De-identified archived data will be stored in a Data Repository. Study source documents (e.g. consent forms, attendance logs) will be retained for up to three years after data analysis is complete. There are no plans to store blood samples for future research. Blood samples drawn for viral load testing will be stored and disposed of according to MOH laboratory procedures.
Supporting Information: Study Protocol, ICF
Time Frame: Once the data is de-identified it may be shared in a repository.
Access Criteria: The team plans to place the data in an open access repository.

REFERENCES:
- [Background] Rahman A, Hamdani SU, Awan NR, Bryant RA, Dawson KS, Khan MF, Azeemi MM, Akhtar P, Nazir H, Chiumento A, Sijbrandij M, Wang D, Farooq S, van Ommeren M. Effect of a Multicomponent Behavioral Intervention in Adults Impaired by Psychological Distress in a Conflict-Affected Area of Pakistan: A Randomized Clinical Trial. JAMA. 2016 Dec 27;316(24):2609-2617. doi: 10.1001/jama.2016.17165. PMID 27837602
- [Background] Bryant RA, Schafer A, Dawson KS, Anjuri D, Mulili C, Ndogoni L, Koyiet P, Sijbrandij M, Ulate J, Harper Shehadeh M, Hadzi-Pavlovic D, van Ommeren M. Effectiveness of a brief behavioural intervention on psychological distress among women with a history of gender-based violence in urban Kenya: A randomised clinical trial. PLoS Med. 2017 Aug 15;14(8):e1002371. doi: 10.1371/journal.pmed.1002371. eCollection 2017 Aug. PMID 28809935
- [Background] Dawson KS, Watts S, Carswell K, Shehadeh MH, Jordans MJD, Bryant RA, Miller KE, Malik A, Brown FL, Servili C, van Ommeren M. Improving access to evidence-based interventions for young adolescents: Early Adolescent Skills for Emotions (EASE). World Psychiatry. 2019 Feb;18(1):105-107. doi: 10.1002/wps.20594. No abstract available. PMID 30600639
- [Background] Epping-Jordan JE, Harris R, Brown FL, Carswell K, Foley C, Garcia-Moreno C, Kogan C, van Ommeren M. Self-Help Plus (SH+): a new WHO stress management package. World Psychiatry. 2016 Oct;15(3):295-296. doi: 10.1002/wps.20355. No abstract available. PMID 27717271
- [Background] Merrill KG, Campbell JC, Decker MR, McGready J, Burke VM, Mwansa JK, Miti S, Frimpong C, Kennedy CE, Denison JA. Prevalence of physical and sexual violence and psychological abuse among adolescents and young adults living with HIV in Zambia. PLoS One. 2020 Jun 25;15(6):e0235203. doi: 10.1371/journal.pone.0235203. eCollection 2020. PMID 32584889
- [Background] Ayano G, Demelash S, Abraha M, Tsegay L. The prevalence of depression among adolescent with HIV/AIDS: a systematic review and meta-analysis. AIDS Res Ther. 2021 Apr 27;18(1):23. doi: 10.1186/s12981-021-00351-1. PMID 33906698
- [Background] Dow DE, Turner EL, Shayo AM, Mmbaga B, Cunningham CK, O'Donnell K. Evaluating mental health difficulties and associated outcomes among HIV-positive adolescents in Tanzania. AIDS Care. 2016 Jul;28(7):825-33. doi: 10.1080/09540121.2016.1139043. Epub 2016 Feb 3. PMID 26837437
- [Background] Boyes ME, Pantelic M, Casale M, Toska E, Newnham E, Cluver LD. Prospective associations between bullying victimisation, internalised stigma, and mental health in South African adolescents living with HIV. J Affect Disord. 2020 Nov 1;276:418-423. doi: 10.1016/j.jad.2020.07.101. Epub 2020 Jul 20. PMID 32871672
- [Background] Pantelic M, Shenderovich Y, Cluver L, Boyes M. Predictors of internalised HIV-related stigma: a systematic review of studies in sub-Saharan Africa. Health Psychol Rev. 2015;9(4):469-90. doi: 10.1080/17437199.2014.996243. Epub 2015 Apr 21. PMID 25559431
- [Background] Pantelic M, Boyes M, Cluver L, Thabeng M. 'They Say HIV is a Punishment from God or from Ancestors': Cross-Cultural Adaptation and Psychometric Assessment of an HIV Stigma Scale for South African Adolescents Living with HIV (ALHIV-SS). Child Indic Res. 2018;11(1):207-223. doi: 10.1007/s12187-016-9428-5. Epub 2016 Nov 23. PMID 29497463
- [Background] Earnshaw VA, Kidman RC, Violari A. Stigma, Depression, and Substance Use Problems Among Perinatally HIV-Infected Youth in South Africa. AIDS Behav. 2018 Dec;22(12):3892-3896. doi: 10.1007/s10461-018-2201-7. PMID 29909588
- [Background] Pantelic M, Boyes M, Cluver L, Meinck F. HIV, violence, blame and shame: pathways of risk to internalized HIV stigma among South African adolescents living with HIV. J Int AIDS Soc. 2017 Aug 21;20(1):21771. doi: 10.7448/IAS.20.1.21771. PMID 28853517
- [Background] Merrill KG, Campbell JC, Decker MR, McGready J, Burke VM, Mwansa JK, Miti S, Frimpong C, Kennedy CE, Denison JA. Past-Year Violence Victimization is Associated with Viral Load Failure Among HIV-Positive Adolescents and Young Adults. AIDS Behav. 2021 May;25(5):1373-1383. doi: 10.1007/s10461-020-02958-3. PMID 32761474
- [Background] Rongkavilit C, Wang B, Naar-King S, Bunupuradah T, Parsons JT, Panthong A, Koken JA, Saengcharnchai P, Phanuphak P. Motivational interviewing targeting risky sex in HIV-positive young Thai men who have sex with men. Arch Sex Behav. 2015 Feb;44(2):329-40. doi: 10.1007/s10508-014-0274-6. Epub 2014 Mar 26. PMID 24668304
- [Background] Pantelic M, Steinert JI, Park J, Mellors S, Murau F. 'Management of a spoiled identity': systematic review of interventions to address self-stigma among people living with and affected by HIV. BMJ Glob Health. 2019 Mar 19;4(2):e001285. doi: 10.1136/bmjgh-2018-001285. eCollection 2019. PMID 30997170
- [Background] Denison JA, Burke VM, Miti S, Nonyane BAS, Frimpong C, Merrill KG, Abrams EA, Mwansa JK. Project YES! Youth Engaging for Success: A randomized controlled trial assessing the impact of a clinic-based peer mentoring program on viral suppression, adherence and internalized stigma among HIV-positive youth (15-24 years) in Ndola, Zambia. PLoS One. 2020 Apr 2;15(4):e0230703. doi: 10.1371/journal.pone.0230703. eCollection 2020. PMID 32240186
- [Background] Andersson GZ, Reinius M, Eriksson LE, Svedhem V, Esfahani FM, Deuba K, Rao D, Lyatuu GW, Giovenco D, Ekstrom AM. Stigma reduction interventions in people living with HIV to improve health-related quality of life. Lancet HIV. 2020 Feb;7(2):e129-e140. doi: 10.1016/S2352-3018(19)30343-1. Epub 2019 Nov 24. PMID 31776098
- [Background] Kalichman S, Mathews C, El-Krab R, Banas E, Kalichman M. Forgoing antiretroviral therapy to evade stigma among people living with HIV, Cape Town, South Africa. J Behav Med. 2021 Oct;44(5):653-661. doi: 10.1007/s10865-021-00212-2. Epub 2021 Mar 31. PMID 33788070
- [Background] Sileo KM, Wanyenze RK, Mukasa B, Musoke W, Kiene SM. The Intersection of Inequitable Gender Norm Endorsement and HIV Stigma: Implications for HIV Care Engagement for Men in Ugandan Fishing Communities. AIDS Behav. 2021 Sep;25(9):2863-2874. doi: 10.1007/s10461-021-03176-1. Epub 2021 Feb 10. PMID 33566214
- [Background] Hargreaves JR, Pliakas T, Hoddinott G, Mainga T, Mubekapi-Musadaidzwa C, Donnell D, Piwowar-Manning E, Agyei Y, Mandla NF, Dunbar R, Macleod D, Floyd S, Bock P, Fidler S, Hayes RJ, Seeley J, Stangl A, Bond V, Ayles H; HPTN 071 (PopART) Study Team. HIV Stigma and Viral Suppression Among People Living With HIV in the Context of Universal Test and Treat: Analysis of Data From the HPTN 071 (PopART) Trial in Zambia and South Africa. J Acquir Immune Defic Syndr. 2020 Dec 15;85(5):561-570. doi: 10.1097/QAI.0000000000002504. PMID 32991336
- [Background] Greenwood GL, Wilson A, Bansal GP, Barnhart C, Barr E, Berzon R, Boyce CA, Elwood W, Gamble-George J, Glenshaw M, Henry R, Iida H, Jenkins RA, Lee S, Malekzadeh A, Morris K, Perrin P, Rice E, Sufian M, Weatherspoon D, Whitaker M, Williams M, Zwerski S, Gaist P. HIV-Related Stigma Research as a Priority at the National Institutes of Health. AIDS Behav. 2022 Jan;26(Suppl 1):5-26. doi: 10.1007/s10461-021-03260-6. Epub 2021 Apr 22. PMID 33886010
- [Background] Scheim AI, Bauer GR. The Intersectional Discrimination Index: Development and validation of measures of self-reported enacted and anticipated discrimination for intercategorical analysis. Soc Sci Med. 2019 Apr;226:225-235. doi: 10.1016/j.socscimed.2018.12.016. Epub 2019 Jan 21. PMID 30674436
- [Background] Fox AB, Earnshaw VA, Taverna EC, Vogt D. Conceptualizing and Measuring Mental Illness Stigma: The Mental Illness Stigma Framework and Critical Review of Measures. Stigma Health. 2018 Nov;3(4):348-376. doi: 10.1037/sah0000104. Epub 2017 Sep 21. PMID 30505939
- [Background] Earnshaw VA, Chaudoir SR. From conceptualizing to measuring HIV stigma: a review of HIV stigma mechanism measures. AIDS Behav. 2009 Dec;13(6):1160-77. doi: 10.1007/s10461-009-9593-3. Epub 2009 Jul 28. PMID 19636699
- [Background] Parker R, Aggleton P. HIV and AIDS-related stigma and discrimination: a conceptual framework and implications for action. Soc Sci Med. 2003 Jul;57(1):13-24. doi: 10.1016/s0277-9536(02)00304-0. PMID 12753813
- [Background] 4. Goffman E. Stigma: Notes on the management of spoiled identity: Simon and Schuster; 2009
- See also: Reference 1 — https://www.unaids.org/sites/default/files/media_asset/2019_women-and-hiv_en.pdf
- See also: Reference 2 — https://www.unicef.org/malawi/media/6266/file/2021%20Global%20Snapshot%20on%20HIV%20&%20AIDS.pdf
- See also: Reference 3 — https://phia.icap.columbia.edu/wp-content/uploads/2019/02/ZAMPHIA-Final-Report__2.22.19.pdf
- See also: Reference 27 — https://www.who.int/publications/i/item/WHO-FWC-MCA-14.05